CLINICAL TRIAL: NCT00510757
Title: Multi Cervical Unit Measures of Cervical Isometric Strength and Range of Motion: A Pilot Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Logan College of Chiropractic (Other)
Responsible Party: Rodger Tepe, PhD, Logan College of Chiropractic
Other Study IDs: RD0426070090
Record Dates: First submitted 2007-07-31; First posted 2007-08-02 (Estimated); Last update posted 2008-10-17 (Estimated); Status verified 2008-10

CONDITIONS: Cervicogenic Headache; Neck Pain; Whiplash; Kyphotic and Reversed Cervical Curves
MeSH Terms: conditions — Post-Traumatic Headache; Neck Pain; Whiplash Injuries

STUDY DESIGN:
Observational Model: Cohort

GROUPS / COHORTS (2):
- Males
- Females

SUMMARY:
This study is designed to collect normative data on cervical isometric strength and range of motion to supplement an existing normative data base.

ELIGIBILITY:
Inclusion Criteria:

* Logan students, faculty and staff

Exclusion Criteria:

* recent surgery,or unstable or fused joints of the cervical spine
* using medications, prescription or herbal muscle stimulants, relaxants, etc
* previous cervical spine injury, surgery or condition that would affect your range of motion in the cervical spine
* currently have any local infection, injury or other malignancy affecting the cervical spine
* congenital conditions affecting the cervical spine, i.e. block vertebrae
* systemic illness with an adverse effect on the cervical spine
* a history of dizziness, light headedness or passing out, or any seizure disorder
* had a neck, shoulder or back injury
* ever been in an automobile accident
* exercise regularly
* pregnant
* spinal manipulation mobilization or other therapy in the last 48 hours

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consenting males and females between the ages of 18 and 65.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2007-06; Primary Completion 2010-06 (Estimated); Study Completion 2010-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Rodger E Tepe, PhD, Principal Investigator — Logan College
Locations (1):
- Logan University, College of Chiropractic, Chesterfield, Missouri, United States